CLINICAL TRIAL: NCT02351648
Title: A Randomised Control Trial of a Transitional Care Model in Singapore General Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Agency for Integrated Care, Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2012/848/E
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Diseases
Keywords: readmission; care transition
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention' (Experimental): Intervention extend from transfer of care to the study team from the initial admission medical team through 90 days after discharge
  Intervention in hospital includes the following. Comprehensive discharge planning based on the 6 principles. Discharge planning initially within 24 hours of recruitment Daily ward review of patients Weekly multi-disciplinary meeting Consolidation of medication and follow-up appointment before discharge Assessment of needs before discharge Comprehensive discharge summary and medication record at discharge
  Intervention after discharge:
  Work done mainly by integrated care nurse Review of patients within 48 hours after discharge via home visit or phone call Subsequent home visit as needed based on patient's needs At least weekly contact with pt or caregiver via telephone Telephone availability working weekday 8 AM to 5 PM Multi-disciplinary meeting for problematic cases Use chronic disease pathway for suitable patients
  Interventions: Other: a transitional care model
- Control' (Active Comparator): Patients receive usual standard of care from the internal medicine team
  Interventions: Other: Control

INTERVENTIONS:
Other: a transitional care model — Intervention extend from transfer of care to the study team from the initial admission medical team through 90 days after discharge
  Intervention in hospital includes the following. Comprehensive discharge planning based on the 6 principles. Discharge planning initially within 24 hours of recruitment Daily ward review of patients Weekly multi-disciplinary meeting Consolidation of medication and follow-up appointment before discharge Assessment of needs before discharge Comprehensive discharge summary and medication record at discharge
  Intervention after discharge:
  Work done mainly by integrated care nurse Review of patients within 48 hours after discharge via home visit or phone call Subsequent home visit as needed based on patient's needs At least weekly contact with pt or caregiver via telephone Telephone availability working weekday 8 AM to 5 PM Multi-disciplinary meeting for problematic cases Use chronic disease pathway for suitable patients
  Arms: Intervention'
Other: Control — Patients receive usual standard of care from the internal medicine team
  Arms: Control'

SUMMARY:
To find out if a transitional care model can reduce the rate of unscheduled readmission to the Department of Internal Medicine (DIM) in SGH

DETAILED DESCRIPTION:
Hospital with high readmission rate is view as having lower quality of care High readmission rate is view as wasteful healthcare spending

Primary Aim:

To find out if a transitional care model can reduce the rate of unscheduled readmission to the Department of Internal Medicine (DIM) in SGH A readmission episode is defined as an episode of readmission to any tertiary hospital within 30 days after index discharge from SGH

Secondary Aim:

To find out if a transitional care model can reduce the number of visits to the emergency department in SGH To find out the quality of our transitional care model by using a care transition measure (CTM-15)

ELIGIBILITY:
Inclusion criteria

-More than 1 admission in the last 90 days

Exclusion Criteria

* Subject is a non-resident
* Subject has no local home address
* Subject is from a long-term care facility during index admission
* Subject is unable to participate in telephone surveillance
* Subject is discharged before takeover
* Subject has impaired decision making capacity without surrogate decision maker
* Subject is pending or currently in critical care unit
* Subject or caregiver is mentally unstable
* Subject is haemodynamically unstable
* Subject requires acute inpatient respiratory support
* Subject requires acute inpatient dialysis support
* Subject pending surgical intervention
* Subject pending transfer to other specialist discipline
* Primary team consultant declined to participate in this research

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Readmission rate | 30 days after index discharge
  A readmission episode is defined as an episode of readmission to any tertiary hospital within 30 days after index discharge from SGH Readmission rate is calculated by dividing the total number of admission by the total number of patients

SECONDARY OUTCOMES:
Readmission rate | up to 180 days after index discharge
  Readmission rate is calculated by dividing the total number of admission by the total number of patients. This will measured at 7 days, 90 days and 180 days of discharge
Quality of transitional care using a validated care transition measure (CTM-15) tool | 90 days after index discharge
  Care transition measure survey of subjects
Emergency department attendance rate | Up to 180 days after index discharge
  Emergency department attendance rate is calculated by dividing the total number of emergency department visits by the total number of patients. This will measured at 7 days, 30 days, 90 days and 180 days of discharge
Time to first readmission | Up to 90 days after index discharge
  Censored time to readmission for both intervention and control group
Specialist Outpatient Clinic visits | Up to 180 days after index discharge
  Outpatient clinic visit rate is calculated by dividing the total number of outpatient clinic visits by the total number of patients. This will measured at 90 days and 180 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kheng Hock Lee, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Coleman EA, Smith JD, Frank JC, Eilertsen TB, Thiare JN, Kramer AM. Development and testing of a measure designed to assess the quality of care transitions. Int J Integr Care. 2002;2:e02. doi: 10.5334/ijic.60. Epub 2002 Jun 1. PMID 16896392
- [Result] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Result] Mistiaen P, Poot E. Telephone follow-up, initiated by a hospital-based health professional, for postdischarge problems in patients discharged from hospital to home. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD004510. doi: 10.1002/14651858.CD004510.pub3. PMID 17054207